CLINICAL TRIAL: NCT05703776
Title: Do Moderately and Severely Depressed Individuals Derive the Same Psychological Benefits From a 10-weeks Long Aerobic Exercise Program ?
Brief Title: Physical Exercise and Depressive Symptoms in Moderately or Severely Depressed Adults
Acronym: EXIMOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Je Bouge Pour Mon Moral (Other)
Collaborators: University Grenoble Alps (Other)
Responsible Party: Principal Investigator, Fabien Legrand, Principal investigator, Je Bouge Pour Mon Moral
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: JBPMM-1
Record Dates: First submitted 2022-10-20; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Depressive Symptoms
Keywords: add-on treatment
MeSH Terms: conditions — Depression | interventions — Nordic Walking

STUDY DESIGN:
Intervention Model Description: open randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nordic Walking (Experimental): 2 weekly sessions of supervised Nordic Walking in a city park with trees, grass, and ponds. Exercise intensity was set at 65%-75% of age-predicted maximal heart rate. The length of training was consecutive 10 weeks
  Interventions: Behavioral: Nordic Walking
- control (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Nordic Walking — Nordic Walking (NW) is an aerobic physical activity where regular walking is enhanced by the addition of the active use of specifically designed NW poles. The physical strain is distributed in a balanced way to various muscle groups of the whole body.
  Arms: Nordic Walking

SUMMARY:
This study is a comparative trial comparing the time course of depressive symptoms between moderately and severely depressed participants over a 10-week long exercise program

DETAILED DESCRIPTION:
Sixty depressed French adults (34 with symptoms of moderate intensity and 26 with symptoms of severe intensity as defined by the PHQ-9 cutting scores) voluntarily participated in our comparative trial.

A control group (waiting list) of n = 16 including 8 severely depressed and 8 moderately depressed participants received no physical exercise.

For the remaining 44 participants (26 with moderate-intensity depressive symptoms and 18 with high-intensity depressive symptoms), two weekly Nordic Walking sessions of 1h were performed for 10 consecutive weeks.

Depressive symptoms were assessed using standard self-report questionnaires at various time points: 1/ enrollment (using the PHQ-9), and then (2) just before the beginning of the exercise intervention (pre-intervention; using the BDI-II), 2/ at the end of Week 5 (mid-intervention; using the BDI-II), and 3/ the day following the end of the exercise program (post-intervention)

ELIGIBILITY:
Inclusion Criteria:

* PHQ-9 (Kroenke et al., 2001) score of 10 or above

Exclusion Criteria:

* medical contraindication to moderate-intensity aerobic exercise
* inability to read French language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
change in the intensity of depressive symptoms | 10 weeks
  self-evaluated intensity of depressive symptoms. Was obtained using the standard Beck Depression Inventory (BDI-II; Beck et al., 1996)

CONTACTS AND LOCATIONS:
Overall Officials: Fabien D Legrand, PhD, Study Director — JBPMM
Locations (1):
- association JBPMM, Nancy, France

IPD SHARING:
Plan to Share IPD: No
Data will be made available upon reasonable request. Requests for access to data from the study should be addressed to Fabien D. Legrand at fabien.legrand@univ-reims.fr. All proposals requesting data access will need to specify how it is planned to use the data, and all proposals will need approval of the study co- investigator team before data release.

REFERENCES:
- [Background] Beck AT, Steer RA, Brown GK. Beck Depression Inventory (2nd edition). San Antonio, TX: Hartcourt Brace, 1996.
- [Background] Kroenke K, Spitzer RL. The PHQ-9: a new depression diagnostic and severity measure. Psychiatric Annals. 2002; 32: 509-521.